CLINICAL TRIAL: NCT00511823
Title: An Open-Label, Three-Part, Two Period, Single Sequence Study to Assess the Pharmacokinetic Interaction Between Repeat Doses of Oral Casopitant and Repeat Oral Doses of Dolasetron, Granisetron or Rosiglitazone When Co-Administered in Healthy Adult Subjects
Brief Title: The Pharmacokinetic Interaction Between Oral Casopitant and Oral Dolasetron, Granisetron or Rosiglitazone in Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKV110483
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: drug-drug interaction,; rosiglitazone,; safety; CYP2C8,; pharmacokinetics,; CYP3A4,; granisetron,; dolasetron,; CYP2D6,; casopitant,
MeSH Terms: conditions — Nausea; Vomiting | interventions — casopitant; dolasetron; Granisetron; Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subjects in Part A (Experimental): Subjects will receive 100 milligrams (mg) of oral dolasetron once daily for 3 days during treatment period 1. In treatment period 2, subjects will receive 100 mg oral dolasetron once daily on days 1, 2 and 3 along with 150 mg oral casopitant on day 1 and 50 mg oral casopitant on days 2 and 3. The treatment periods will be separated by will be separated by a 5 - 14 day wash-out period.
  Interventions: Drug: casopitant; Drug: dolasetron
- Subjects in Part B (Experimental): Subjects will receive 2 mg of oral granisetron once daily for 3 days during treatment period 1. In treatment period 2, subjects will receive 2 mg oral granisetron once daily on days 1, 2 and 3 along with 150 mg oral casopitant once daily on day 1 and 50 mg oral casopitant once daily on days 2 and 3. The treatment periods will be separated by will be separated by a 5 - 14 day wash-out period.
  Interventions: Drug: casopitant; Drug: granisetron
- Subjects in Part C (Experimental): Subjects will receive 4 mg of oral rosiglitazone once daily for 3 days during treatment period 1. In treatment period 2, subjects will receive 4 mg oral rosiglitazone once daily on days 1, 2 and 3 along with 150 mg oral casopitant once daily on day 1 and 50 mg oral casopitant once daily on days 2 and 3. The treatment periods will be separated by will be separated by a 5 - 14 day wash-out period.
  Interventions: Drug: casopitant; Drug: rosiglitazone

INTERVENTIONS:
Drug: casopitant — The doses of casopitant will be comprised of 150 mg (one 150 mg tablet) and 50 mg (one 50 mg tablet). Casopitant will be taken with 240 milliliters (mL) of water on an empty stomach following at least 2 hour fast.
Drug: dolasetron — The dose of oral dolasetron will be comprised of 100 mg (one 100 mg tablet or two 50 mg tablets). Dolasetron will be taken with 240 mL of water on an empty stomach following at least 2 hour fast.
  Arms: Subjects in Part A
Drug: granisetron — The dose of oral granisetron will be comprised of 2 mg (two 1 mg tablets). Granisetron will be taken with 240 mL of water on an empty stomach following at least 2 hour fast.
  Arms: Subjects in Part B
Drug: rosiglitazone — The dose of oral rosiglitazone will be comprised of 4 mg (two 2 mg tablets or one 4 mg tablet). Rosiglitazone will be taken with 240 mL of water on an empty stomach following at least 2 hour fast.
  Arms: Subjects in Part C

SUMMARY:
This A Three-Part Drug-Drug Interaction Study To Evaluate Effects of Casopitant On Dolasetron, Granisetron or Rosiglitazone When Co-Administered in Healthy Adults

ELIGIBILITY:
Inclusion Criteria:

* An adult healthy male or female.
* Age: 18 to 64 years, inclusive.
* Body mass index (BMI) = 19 to = 37 kg/m2.
* A female if she is of Non-childbearing potential, OR
* A female who has a negative serum pregnancy test within 14 days prior to the first dose of study medication and agrees to use adequate contraception during the study and for 14 days after the last dose of study medication.
* Adequate organ systems function [Hemoglobin is within normal limits ± 10%; Platelets is = 100 X 109/L or = lower limit of normal (LLN); Aspartate aminotransaminase = Upper limit of normal (ULN); Total bilirubin = 1.2 times ULN; Creatine phosphokinase < 1.5 times ULN; Renal Calculated creatinine clearance = 50 mL/min]
* Able to swallow and retain oral medication.
* Able to understand and comply with the requirements, instruction and restrictions stated in the informed consent.
* Signed and dated informed consent.

Exclusion Criteria:

* Clinically relevant abnormality, including any degree of heart failure or clinically significant cardiac disease, identified on the screening exam or any other medical condition or circumstance making the subject unsuitable for participation in the study.
* For Part A (dolasetron-casopitant drug-drug interaction), any subject who exhibits gene duplication for CYP2D6.
* History of drug or other allergy which, in the opinion of the Investigator, contraindicates participation.
* Known immediate hypersensitivity reaction or idiosyncrasy to study drugs or any drug chemically related to the study medications.
* Use of an investigational drug within 28 days or 5 half-lives, whichever is longer, preceding the first dose of study medication(s).
* Blood donation in excess of 500 mL within 56 days prior to dosing or intends to donate within 30 days of the post-treatment follow-up visit.
* Presence of or suspected iron deficiency.
* Stool positive for occult blood.
* Troponin I level above 10% of the coefficient of variation of the assay.
* For female subjects of childbearing potential, a positive serum pregnancy test.
* Female subject who is lactating.
* Positive urine drug screen (UDS) including alcohol.
* Positive for HIV antibody, hepatitis C antibody or hepatitis B surface antigen (HBsAg).
* Positive urinary cotinine.
* Smoking history of = 4 packs per day/year or smoked more than 2 times within the past 30 days prior to screening.
* History of drug abuse or dependence within 6 months of screening.
* History of alcohol abuse within 6 months of screening or alcohol consumption in the past 6 months exceeding 7 drinks/week for women and 14 drinks/week for men (where 1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor).
* Presence of an active infection.
* Corrected QT interval (QTc) > 450 msecs.
* Pepsinogen level below the lower limit of laboratory reference range (LLRR).
* Active peptic ulcer disease (PUD) or a history of PUD of unknown etiology.
* Use of any prescription or non-prescription drug(s), including oral contraceptives, herbal or dietary supplements or vitamins within 14 days, or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Consumption of food or drink containing grapefruit or grapefruit juice, apple juice, Seville oranges, kumquats, pomelos, star fruit, red wine, charbroiled meats, cabbage or vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard) within 7 days prior to the first dose of study medication(s).
* History of cholecystectomy or biliary tract disease.
* Any serious or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-07-23 (Actual); Primary Completion 2007-09-21 (Actual); Study Completion 2007-09-21 (Actual)

PRIMARY OUTCOMES:
Change of AUC and Cmax of dolasetron, granisetron and rosiglitazone after oral administration alone and co-administered with oral casopitant | (comparing AUC & Cmax of Days 1&3 of the Period One and Two)

SECONDARY OUTCOMES:
Safety evaluations of AEs and changes in laboratory values, ECGs, vitals evaluated during the study | (Day -1 and Days 1-4 of the Period One and Two, at follow-up visit)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Adams LM, Johnson B, Zhang K, Yue L, Kirby LC, Lebowitz P, Stoltz R. Effect of casopitant, a novel NK-1 antagonist, on the pharmacokinetics of dolasetron and granisetron. Support Care Cancer. 2009 Sep;17(9):1187-93. doi: 10.1007/s00520-008-0572-4. Epub 2009 Feb 10. PMID 19205754
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study NKV110483 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/NKV110483?search=study&search_terms=NKV110483#rs
- Available data/document: Clinical Study Report: NKV110483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKV110483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKV110483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKV110483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKV110483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKV110483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKV110483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register